CLINICAL TRIAL: NCT02329665
Title: A Prospective Data Collection, Single-Center, Open Label Study in Patients Undergoing CT-Guided Needle Interventions for the Development of the NeedleWays System
Brief Title: Data Collection in Patients Undergoing CT-Guided Needle Interventions for NeedleWays System Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeedleWays (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NW-CL-001P-IL
Record Dates: First submitted 2014-12-20; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeedleWays™ System (Experimental): A total of 50 consecutive subjects scheduled for clinically indicated CT guided needle intervention procedure will be invited to enroll in the study.
  Interventions: Device: NeedleWays™ System

INTERVENTIONS:
Device: NeedleWays™ System — A total of 50 consecutive subjects scheduled for clinically indicated CT guided needle intervention procedure will be invited to enroll in the study.

SUMMARY:
The primary objective of this study is to collect CT images of patients undergoing CT Guided Needle Intervention Procedures which will be used for the development of the NeedleWaysTM System.

DETAILED DESCRIPTION:
The study will collect anonymized data in support of further development of the NeedleWays System.

The collected data will be:

1. Anonymized CT scans with Patient Reference Frame (PRF) placed upon the scanned area, outside of the sterile field.
2. Screen captures of the NeedleWays Procedure console display as the intervention needle is placed on the patients body, outside of the sterile field.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects, 18 years of age or older at the time of enrollment.
* Subjects meeting all medical conditions for percutaneous CT-guided needle intervention.
* INR <1.4
* Written informed consent to participate in the study.
* Ability to comply with the requirements of the study procedures. Exclusion Criteria
* Subjects diagnosed with one or more of the following according to medical records:
* Hemophilia, thrombocytopenia, coagulopathy, or other elevated risk for bleeding or abnormal clotting,Pulmonary hypertension, heart failure, renal failure, or blood dyscrasia
* Subjects treated with Ticlopidine or similar antithrombotic medication.
* Subjects who cannot tolerate mild sedation
* Subjects with the following laboratory values, unless otherwise approved by hematologist:
* Platelet count <60,000/ml
* APTT >39 sec or PT >15 sec
* Pregnancy or lactation
* Subject is unable to comply with requirements of the procedure, i.e. holding breath.
* Subject participation in an investigational trial within 30 days of enrollment
* Subjects who are uncooperative or cannot follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
collect CT images of patients undergoing CT | procedure duration
  The primary objective of this study is to collect CT images of patients undergoing CT Guided Needle Intervention Procedures which will be used for the development of the NeedleWaysTM System.